CLINICAL TRIAL: NCT06368232
Title: Evaluation Of Nutritional Status Of Morbid Obesity Patients In The First Six Months After Sleeve Gastrectomy
Brief Title: Nutritional Status After Sleeve Gastrectomy in Morbid Obesity: 6-Month Study
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assistant Professor, Ankara Yildirim Beyazıt University
Other Study IDs: 19.036.123.125
Record Dates: First submitted 2024-03-26; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Bariatric Surgery Candidate; Gastrostomy; Obesity
Keywords: Gastrectomy; Bariatric Surgery; Nutritional Status
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: püPatients undergoing bariatric surgery — Patients will not be intervened. Only nutritional status after bariatric surgery will be evaluated.The data of 76 patients aged 19-64 years who had undergone bariatric surgery and were followed by a dietitian dietitian for at least 6 months were included.

SUMMARY:
This study aims to evaluate the nutritional status of morbidly obese patients following gastric bypass surgery. Data from 76 patients aged 19-64, who will be monitored by a dietitian for at least six months, will be analyzed. Preoperative and postoperative biochemical parameters along with anthropometric measurements will assess.

DETAILED DESCRIPTION:
Objective: This retrospective study aims to evaluate the nutritional status of morbidly obese patients in the first six months following sleeve gastrectomy.

Methods: The study is planned as a retrospective analysis. The data of 76 patients aged 19-64 years who underwent bariatric surgery and were monitored by a dietitian for at least six months will be included in the study. Preoperative and postoperative biochemical parameters and anthropometric measurements of the patients will be collected and analyzed.

Detailed Description: The study will assess the changes in nutritional status, including body weight, BMI, fasting blood glucose, HbA1c, Homa-IR, iron levels, vitamin D levels, and lipid profile (triglycerides, LDL, HDL) among morbidly obese patients in the first six months following sleeve gastrectomy. Preoperative and postoperative measurements will be compared to evaluate the impact of surgery on these parameters.

Conclusion: Results will be analyzed and interpreted after data collection is completed, and conclusions will be drawn accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Data of patients aged 19-64 years
* Data of patients with BMI ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 and at least one comorbidity such as obesity-related hypertension, dyslipidemia, type 2 diabetes mellitus, and sleep apnea
* Data of patients who underwent sleeve gastrectomy
* Volunteering

Exclusion Criteria:

* Data of patients who were not deemed suitable for surgery by the physician and to whom a surgical technique different from sleeve gastrectomy was applied
* Data of patients who were not followed up by a dietitian for six months after surgery
* Data of patients with gastrointestinal inflammatory bowel disease
* Data of patients with psychiatric disorders diagnosed by a physician
* Data of patients with cancer, pregnant and lactating women, alcohol or drug addiction

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Data from 76 patients aged 19-64 years who applied to the General Surgery Obesity and Metabolic Surgery clinic and were followed up for six months were included.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Body Weight | Preoperative period, postoperative months 1 and 6
  Kilograms (kg)
BMI (Body Mass Index) | Preoperative period, postoperative months 1 and 6
  Kilograms per square meter (kg/m2)
Lean Mass | Preoperative period, postoperative months 1 and 6
  Kilograms (kg)
Fat Mass | Preoperative period, postoperative months 1 and 6
  Kilograms (kg)
Fasting Blood Glucose | Preoperative period, postoperative months 1 and 6
  Milligrams per deciliter (mg/dL)
HbA1c | Preoperative period, postoperative months 1 and 6
  Percentage (%)
Iron levels | Preoperative period, postoperative months 1 and 6
  Micrograms per deciliter (µg/dL)
Vitamin D level | Preoperative period, postoperative months 1 and 6
  Nanograms per milliliter (ng/mL)
Lipid Profile (Triglycerides, LDL, HDL) | Preoperative period, postoperative months 1 and 6
  Milligrams per deciliter (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Yahya Özdoğan, Assoc. Prof, Principal Investigator — Ankara Yıldırım Beyazıt Üniversity
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) don't be available to other researchers